CLINICAL TRIAL: NCT04907227
Title: A Phase 3, Randomized, Double-blind Study of Pembrolizumab (MK-3475) Plus Docetaxel Plus Prednisone Versus Placebo Plus Docetaxel Plus Prednisone in Participants With Chemotherapy-naïve Metastatic Castration-Resistant Prostate Cancer (mCRPC) Who Have Progressed on a Next Generation Hormonal Agent (NHA) (KEYNOTE-921)
Brief Title: Study of Pembrolizumab (MK-3475) Plus Docetaxel Versus Placebo Plus Docetaxel in Chemotherapy-naïve Metastatic Castration-resistant Prostate Cancer (mCRPC) (MK-3475-921/KEYNOTE-921)-China Extension
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The data did not support study endpoints
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3475-921 China Extension; MK-3475-921 China Extension (Other: Merck); KEYNOTE-921 (Other: Merck); 194831 (Registry Identifier: JAPAC-CTI)
Record Dates: First submitted 2021-05-26; First posted 2021-05-28 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: Prostatic Neoplasms
Keywords: Programmed Cell Death 1 (PD 1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL 1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL 2, PD-L2)
MeSH Terms: conditions — Prostatic Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Docetaxel; Prednisone; Saline Solution; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pembrolizumab+Docetaxel (Experimental): Participants receive pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W) for up to a maximum of 35 cycles (approximately 2 years) PLUS docetaxel 75 mg/m^2 by IV infusion on Day 1 of each 21-day cycle (Q3W) for a maximum of 10 cycles (approximately 7 months). Participants also concomitantly receive dexamethasone 8 mg by oral tablets at 12 hours, 3 hours, and 1 hour prior to docetaxel administration and prednisone 5 mg by oral tablets twice daily during each 21-day docetaxel cycle.
  Interventions: Biological: Pembrolizumab; Drug: Docetaxel; Drug: Prednisone; Drug: Dexamethasone
- Placebo+Docetaxel (Placebo Comparator): Participants receive placebo by IV infusion on Day 1 of each 21-day cycle (Q3W) for up to a maximum of 35 cycles (approximately 2 years) PLUS docetaxel 75 mg/m^2 by IV infusion on Day 1 of each 21-day cycle (Q3W) for a maximum of 10 cycles (approximately 7 months). Participants also concomitantly receive dexamethasone 8 mg by oral tablets at 12 hours, 3 hours, and 1 hour prior to docetaxel administration and prednisone 5 mg by oral tablets twice daily during each 21-day docetaxel cycle.
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: Placebo; Drug: Dexamethasone

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab+Docetaxel
Drug: Docetaxel — IV infusion
  Other Names: TAXOTERE®
Drug: Prednisone — Oral tablets
Drug: Placebo — IV infusion
  Other Names: Normal saline or dextrose infusion
  Arms: Placebo+Docetaxel
Drug: Dexamethasone — Oral tablets
  Other Names: DECADRON®

SUMMARY:
The purpose of this study is to assess the efficacy and safety of the combination of pembrolizumab (MK-3475) and docetaxel in the treatment of Chinese men with metastatic castration-resistant prostate cancer (mCRPC) who have not received chemotherapy for mCRPC but have progressed on or are intolerant to Next Generation Hormonal Agent (NHA).

There are two primary study hypotheses.

Hypothesis 1: The combination of pembrolizumab plus docetaxel plus prednisone is superior to placebo plus docetaxel plus prednisone with respect to Overall Survival (OS).

Hypothesis 2: The combination of pembrolizumab plus docetaxel plus prednisone is superior to placebo plus docetaxel plus prednisone with respect to Radiographic Progression-free Survival (rPFS) per Prostate Cancer Working Group (PCWG)-modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by blinded independent central review.

DETAILED DESCRIPTION:
The China extension study will include participants previously enrolled in China in the global study for MK-3475-921 (NCT03834506) plus those enrolled during the China extension enrollment period.

With Amendment 6 (effective date: 29-Sep-2022), all participants were unblinded and placebo treatment was stopped. Participants deemed to derive clinical benefit from treatment may have continued at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically- or cytologically-confirmed adenocarcinoma of the prostate without small cell histology
* Has prostate cancer progression while on androgen deprivation therapy (or post bilateral orchiectomy) within 6 months prior to screening
* Has current evidence of metastatic disease documented by either bone lesions on bone scan and/or soft tissue disease by computed tomography/magnetic resonance imaging (CT/MRI)
* Has received prior treatment with one (but not more than one) NHA (eg, abiraterone acetate, enzalutamide, apalutamide, or darolutamide) for metastatic hormone-sensitive prostate cancer (mHSPC) or castration-resistant prostate cancer (CRPC) and either a) progressed through treatment OR b) has become intolerant of the drug
* Has ongoing androgen deprivation with serum testosterone <50 ng/dL (<2.0 nM)
* Participants receiving bone resorptive therapy (including, but not limited to, bisphosphonate or denosumab) must have been on stable doses prior to randomization
* Participants must agree to the following during the study treatment period and for at least 120 days after the last dose of pembrolizumab or for at least 180 days after the last dose of docetaxel (whichever is longer): Refrain from donating sperm PLUS Use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause)
* Participants must agree to use male condom when engaging in any activity that allows for passage of ejaculate to another person of any sex
* Has provided newly obtained core or excisional biopsy (obtained within 12 months of screening) from soft tissue not previously irradiated (samples from tumors progressing in a prior site of radiation are allowed). Participants with bone only or bone predominant disease may provide a bone biopsy sample
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 assessed within 7 days of randomization

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active treatment in the last 3 years
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy
* Has undergone major surgery including local prostate intervention (excluding prostate biopsy) within 28 days prior to randomization and not recovered adequately from the toxicities and/or complications
* Has a gastrointestinal disorder affecting absorption or is unable to swallow tablets/capsules
* Has an active infection (including tuberculosis) requiring systemic therapy
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has known active human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients
* Has symptomatic congestive heart failure (New York Heart Association Class III or IV heart disease)
* Has had a prior anti-cancer monoclonal antibody (mAb) prior to randomization or who has not recovered (i.e., Grade ≤1 or at baseline) from AEs due to mAbs
* Has used herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA levels (e.g. saw palmetto) prior to randomization
* Has received prior treatment with radium or other therapeutic radiopharmaceuticals for prostate cancer
* Has received prior therapy with an anti-programmed cell death-1 (anti-PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1), or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX-40, CD137)
* Has received prior treatment with docetaxel or another chemotherapy agent for mCRPC
* Has hypersensitivity to docetaxel or polysorbate 80
* Is currently receiving either strong or moderate inhibitors of cytochrome P450 (CYP)3A4 that cannot be discontinued for the duration of the study
* Has received prior targeted small molecule therapy or abiraterone acetate, enzalutamide, apalutamide, or darolutamide within 4 weeks prior to the first dose of study treatment, or has not recovered (i.e., Grade ≤1 or at baseline) from AEs due to a previously administered agent
* Has received prior radiotherapy to within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis
* Has received a live vaccine within 30 days prior to randomization
* Has received treatment with 5α reductase inhibitors (eg, finasteride or dutasteride), estrogens, and/or cyproterone within 4 weeks prior to randomization
* Has received prior treatment with ketoconazole for prostate cancer
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Has a "superscan" bone scan
* Is expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2023-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (20):
- China (20):
  - Second Affiliated hospital of Anhui Medical University-Urology (Site 1339), Hefei, Anhui
  - Peking University First Hospital ( Site 1303), Beijing, Beijing Municipality
  - The Fifth Medical Center of PLA General Hospital ( Site 1307), Beijing, Beijing Municipality
  - Peking University Third Hospital (Site 1304), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 1305), Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University ( Site 1319), Xiamen, Fujian
  - Sun Yat Sen Memorial Hospital ( Site 1323), Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University ( Site 1330), Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center (Site 1334), Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital (Site 1326), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 1321), Zhengzhou, Henan
  - Hubei Cancer Hospital ( Site 1329), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 1320), Changsha, Hunan
  - Nanjing Drum Tower Hospital ( Site 1312), Nanjing, Jiangsu
  - Zhongshan Hospital Fudan University ( Site 1301), Shanghai, Shanghai Municipality
  - Renji Hospital Shanghai Jiao Tong University School of Medicine (Site 1335), Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center ( Site 1300), Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi an Jiaotong University (Site 1315), Xian, Shanxi
  - The Second Affiliated Hospital of Zhejiang University School of Medicine ( Site 1309), Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital ( Site 1310), Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol-specified final analysis for all primary and secondary outcome measures was performed with the primary completion data cutoff.
  Twenty-one participants in the China extension study were also included in the global study for MK-3475-921 (NCT03834506).
Groups:
- Pembrolizumab + Docetaxel: Participants received pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W) for up to a maximum of 35 cycles (approximately 2 years) PLUS docetaxel 75 mg/m^2 by IV infusion on Day 1 of each 21-day cycle (Q3W) for a maximum of 10 cycles (approximately 7 months). Participants also concomitantly received dexamethasone 8 mg by oral tablets at 12 hours, 3 hours, and 1 hour prior to docetaxel administration and prednisone 5 mg by oral tablets twice daily during each 21-day docetaxel cycle.
- Placebo + Docetaxel: Participants received placebo by IV infusion on Day 1 of each 21-day cycle (Q3W) for up to a maximum of 35 cycles (approximately 2 years) PLUS docetaxel 75 mg/m^2 by IV infusion on Day 1 of each 21-day cycle (Q3W) for a maximum of 10 cycles (approximately 7 months). Participants also concomitantly received dexamethasone 8 mg by oral tablets at 12 hours, 3 hours, and 1 hour prior to docetaxel administration and prednisone 5 mg by oral tablets twice daily during each 21-day docetaxel cycle.
Period: Overall Study
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Started | 41 | 40
Treated | 41 | 40
Completed | 0 | 0
Not Completed | 41 | 40
Not completed — Death | 12 | 8
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Withdrawal By Parent/Guardian | 1 | 0
Not completed — Sponsor Decision | 25 | 30
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.1 (7.5) | 68.0 (7.5) | 67.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 41 | 40 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 40 | 39 | 79
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 41 | 40 | 81
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. The OS was calculated using the product-limit Kaplan-Meier (K-M) method for censored data. Participants without documented death at the time of the analysis were censored at the date of the last follow-up. Per protocol, final analysis for this outcome measure was performed with the primary completion data cutoff.
Time Frame: Up to 19.8 months
Population: All randomized participants in the intent to treat population who had data available for analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 41 | 40
Months | 16.3 [10.6 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 13.9 [11.1 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Docetaxel vs Placebo + Docetaxel; Test type: Other; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.32 to 2.46] — HR based on Cox regression model with Efron's method of tie handling with treatment as a covariate

2. Primary Outcome: Radiographic Progression-free Survival (rPFS) Per Prostate Cancer Working Group (PCWG)-Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: rPFS was defined as the time from randomization to occurrence of: radiological tumor progression using RECIST 1.1 as assessed by BICR; progression of bone lesions using PCWG criteria; or death due to any cause. Radiological progression as per RECIST 1.1 was ≥20% increase in sum of diameters of target lesions and progression of existing non-target lesions. Progression of bone lesions by PCWG criteria was the appearance of ≥2 new bone lesions on bone scan, that have been confirmed to not represent tumor flare, and was persistent for ≥6 weeks. The rPFS was calculated using the product-limit K-M method for censored data. Participants without a rPFS event were censored at the date of last disease assessment. Per protocol, final analysis for this outcome measure was performed with the primary completion data cutoff.
Time Frame: Up to 19.8 months
Population: All randomized participants in the intent to treat population who had data available for analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 41 | 40
Months | 6.4 [4.2 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 11.2 [6.3 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Docetaxel vs Placebo + Docetaxel; Test type: Other; Hazard Ratio (HR) = 1.59, 95% CI 2-sided [0.68 to 3.67] — HR based on Cox regression model with Efron's method of tie handling with treatment as a covariate

3. Secondary Outcome: Time to Initiation of the First Subsequent Anti-cancer Therapy (TFST)
Description: TFST was defined as the time from randomization to initiation of the first subsequent anti-cancer therapy or death; whichever occurred first. The TFST was calculated using the product-limit K-M method for censored data. Any participant not known to have further subsequent therapy or death was censored at the last known time that no subsequent new anti-cancer therapy was received. Per protocol, final analysis for this outcome measure was performed with the primary completion data cutoff.
Time Frame: Up to 19.8 months
Population: All randomized participants in the intent to treat population who had data available for analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 41 | 40
Months | 9.3 [5.8 to 10.1] | 8.3 [4.9 to 10.2]
Statistical Analysis 1: Comparison: Pembrolizumab + Docetaxel vs Placebo + Docetaxel; Test type: Other; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.45 to 1.50] — HR based on Cox regression model with Efron's method of tie handling with treatment as a covariate

4. Secondary Outcome: Prostate-specific Antigen (PSA) Response Rate
Description: The Prostate-specific Antigen (PSA) response rate was the percentage of participants who had PSA response defined as a reduction in the PSA level from baseline by ≥50%. The reduction in PSA level was confirmed by an additional PSA evaluation performed ≥3 weeks from the original response. The analysis was performed on participants who had baseline PSA measurements. Per protocol, final analysis for this outcome measure was performed with the primary completion data cutoff.
Time Frame: Up to 19.8 months
Population: All randomized participants in the intent to treat population, who had a PSA measurement at baseline, and had data available for analysis
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 41 | 40
Percentage of participants | 24.4 [12.4 to 40.3] | 22.5 [10.8 to 38.5]

5. Secondary Outcome: Objective Response Rate (ORR) Per Prostate Cancer Working Group (PCWG)-Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: ORR was defined as the percentage of participants with complete response (CR: disappearance of all target lesions per RECIST 1.1; and no evidence of disease (NED) on bone scan per PCWG) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions per RECIST 1.1; and non-progressive disease, non-evaluable [NE], or NED on bone scan or CR with non-progressive disease or NE bone scan per PCWG). Per protocol, final analysis for this outcome measure was performed with the primary completion data cutoff.
Time Frame: Up to 19.8 months
Population: All randomized participants in the intent to treat population, with measurable disease at baseline, and had data available for analysis
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 17 | 15
Percentage of participants | 17.6 [3.8 to 43.4] | 13.3 [1.7 to 40.5]
Statistical Analysis 1: Comparison: Pembrolizumab + Docetaxel vs Placebo + Docetaxel; Test type: Other; Percent Difference = 4.3, 95% CI 2-sided [-24.1 to 31.2] — Based on Miettinen & Nurminen method

6. Secondary Outcome: Duration of Response (DOR) Per Prostate Cancer Working Group (PCWG)-Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: DOR was the time from first evidence of complete response (CR: disappearance of all target lesions per RECIST 1.1; and no evidence of disease [NED] on bone scan per PCWG) or partial response (PR: ≥30% decrease in the sum of diameters of target lesions per RECIST 1.1; non-progressive disease, non-evaluable [NE], or NED on bone scan or CR with non-progressive disease or NE bone scan per PCWG) until progressive disease (PD) or death. PD per RECIST 1.1 was ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. PD per PCWG was the appearance of ≥2 new bone lesions on bone scan that were confirmed to not represent tumor flare and persisted for ≥6 weeks. DOR was calculated using the product-limit K-M method. Participants who did not progress were censored at last disease assessment. Per protocol final analysis for this outcome measure was done with the primary completion data cutoff.
Time Frame: Up to 19.8 months
Population: All randomized participants in the intent to treat population, who demonstrated a CR or PR, and had data available for analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 3 | 2
Months | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of responding participants with relapse.

7. Secondary Outcome: Time to Pain Progression (TTPP) as Assessed by Brief Pain Inventory-Short Form (BPI-SF) Item 3 ("Worst Pain in 24 Hours") and Opiate Analgesic Use Assessed by the Analgesic Quantification Algorithm [AQA] Score
Description: TTPP was time from randomization to pain progression (PP) per BPI-SF Item 3 and AQA score. BPI-SF assesses pain intensity; for item 3, responses to "Please rate your pain at its worst in the last 24 hours" are scored from 0 (no pain) to 10 (worst pain). A higher score indicates greater pain. AQA captures the intensity of analgesic use, scored from 0 (no use) to 7 (strong opioid use). A higher score indicates higher intensity of use.
  For participants asymptomatic at baseline, PP was ≥2-point change from baseline in Item 3 score OR opioid use initiation. For those symptomatic at baseline, PP was ≥2-point change from baseline in Item 3 score, a score of ≥4, no decrease in average opioid use OR any increase in opioid use (e.g. 1 point change in AQA score). TTPP was assessed by product-limit K-M method. Participants with >2 consecutive unevaluable visits were censored at last assessment. Per protocol final analysis for this outcome measure was done with the primary completion data cutoff.
Time Frame: Up to 19.8 months
Population: All participants in the participant-reported outcomes (PRO) full analysis set who received ≥1 dose of study treatment and who had ≥1 PRO assessment available
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 41 | 40
Months | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Docetaxel vs Placebo + Docetaxel; Test type: Other; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.17 to 1.99] — HR based on Cox regression model with Efron's method of tie handling with treatment as a covariate

8. Secondary Outcome: Time to First Symptomatic Skeletal-related Event (SSRE)
Description: SSRE was the time from randomization to the first symptomatic skeletal-related event defined as: 1. use of external-beam radiation therapy (EBRT) to prevent or relieve skeletal symptoms 2. occurrence of new symptomatic pathologic bone fracture (vertebral or non-vertebral) 3. occurrence of spinal cord compression 4. tumor-related orthopedic surgical intervention, whichever occurs first. The SSRE was calculated using the product-limit K-M method for censored data. Participants without symptomatic skeletal-related events were censored at the last evaluable assessment. Per protocol, final analysis for this outcome measure was performed with the primary completion data cutoff.
Time Frame: Up to 19.8 months
Population: All randomized participants in the intent to treat population who had data available for analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 41 | 40
Months | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [10.0 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Docetaxel vs Placebo + Docetaxel; Test type: Other; Hazard Ratio (HR) = 1.64, 95% CI 2-sided [0.15 to 18.24] — HR based on Cox regression model with Efron's method of tie handling with treatment as a covariate

9. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: The time to PSA progression was the time from randomization to PSA progression. The PSA progression date was defined as the date of: 1. ≥25% increase and ≥2 ng/mL above the nadir, confirmed by a second value ≥3 weeks later if there was PSA decline from baseline; OR 2. ≥25% increase and ≥2 ng/mL increase from baseline beyond 12 weeks if there was no PSA decline from baseline. Time to PSA progression was calculated using the product-limit K-M method for censored data. Participants without PSA progression were censored at the last evaluable assessment. Per protocol, final analysis for this outcome measure was performed with the primary completion data cutoff.
Time Frame: Up to 19.8 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 41 | 40
Months | 5.0 [3.0 to 9.6] | 3.7 [2.8 to 6.7]
Statistical Analysis 1: Comparison: Pembrolizumab + Docetaxel vs Placebo + Docetaxel; Test type: Other; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.41 to 1.46] — HR based on Cox regression model with Efron's method of tie handling with treatment as a covariate

10. Secondary Outcome: Time to Radiographic Soft Tissue Progression Per Soft Tissue Rules of Prostate Cancer Working Group (PCWG)-Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: The time to radiographic soft tissue progression was defined as the time from randomization to radiographic soft tissue progression per soft tissue rules of PCWG-modified RECIST 1.1 as assessed by BICR. Progression was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered progression. Time to radiographic soft tissue progression was calculated using the product-limit K-M method for censored data. Participants without radiographic soft tissue progression were censored at the last evaluable assessment. Per protocol, final analysis for this outcome measure was performed with the primary completion data cutoff.
Time Frame: Up to 19.8 months
Population: All randomized participants in the intent to treat population who had data available for analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 41 | 40
Months | NA [8.2 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 11.2 [8.2 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Docetaxel vs Placebo + Docetaxel; Test type: Other; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.43 to 3.17] — HR based on Cox regression model with Efron's method of tie handling with treatment as a covariate

11. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Per protocol, final analysis for this outcome measure was performed with the primary completion data cutoff. The number of participants who experienced an AE is presented.
Time Frame: Up to 17 months
Population: All participants who received ≥1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 41 | 40
Participants | 37 | 34

12. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due To an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Per protocol, final analysis for this outcome measure was performed with the primary completion data cutoff. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to 14 months
Population: All participants who received ≥1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 41 | 40
Participants | 3 | 6

ADVERSE EVENTS:
Time Frame: Up to approximately 31 months
Description: All-cause mortality: All randomized participants; AEs: all participants who received ≥1 dose of study treatment. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study drug. Therefore, Medical Dictionary for Regulatory Activities (MedDRA) preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
All-Cause Mortality (participants affected / at risk) | 12/41 | 9/40
Serious Adverse Events (participants affected / at risk) | 11/41 | 12/40
Other Adverse Events (participants affected / at risk) | 36/41 | 34/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Docetaxel (N=41) | Placebo + Docetaxel (N=40)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation proctitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (3)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Docetaxel (N=41) | Placebo + Docetaxel (N=40)
Anaemia (Blood and lymphatic system disorders) | 23 (36) | 20 (52)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 8 (12) | 9 (11)
Diarrhoea (Gastrointestinal disorders) | 5 (8) | 5 (7)
Nausea (Gastrointestinal disorders) | 3 (3) | 6 (8)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Asthenia (General disorders) | 5 (13) | 5 (5)
Chest discomfort (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 7 (11) | 3 (3)
Malaise (General disorders) | 2 (4) | 4 (7)
Oedema peripheral (General disorders) | 5 (5) | 4 (5)
Pain (General disorders) | 2 (2) | 3 (4)
Pyrexia (General disorders) | 3 (3) | 6 (8)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 3 (3)
Alanine aminotransferase increased (Investigations) | 3 (5) | 4 (7)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (8)
Blood alkaline phosphatase increased (Investigations) | 3 (5) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (7) | 5 (18)
Neutrophil count decreased (Investigations) | 12 (40) | 18 (53)
Platelet count decreased (Investigations) | 5 (11) | 5 (5)
Tri-iodothyronine decreased (Investigations) | 1 (1) | 3 (3)
Weight decreased (Investigations) | 4 (4) | 5 (5)
White blood cell count decreased (Investigations) | 20 (53) | 18 (63)
White blood cell count increased (Investigations) | 2 (4) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 8 (10) | 10 (14)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 (5) | 4 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 4 (5)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (6) | 3 (8)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (13)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 7 (13)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (11) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1) | 4 (4)
Proteinuria (Renal and urinary disorders) | 3 (4) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10) | 11 (12)
Nail discolouration (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (10) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (7) | 6 (9)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT04907227/Prot_SAP_000.pdf